CLINICAL TRIAL: NCT02580799
Title: Immunohistochemical HER2 Status Evaluation In Breast Cancer Pathology Samples: A Multicenter, Parallel-Design Concordance Study
Brief Title: Study of Human Epidermal Growth Receptor (HER2) Status Evaluation in Breast Cancer Pathology Samples
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28731
Record Dates: First submitted 2015-10-19; First posted 2015-10-20 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast Cancer Pathology Samples: Breast cancer pathology samples were evaluated for a period of 70 days.

SUMMARY:
A multi-center non-interventional, in-vitro trial for evaluation of concordance of the results for Human Epidermal Growth Factor Receptor 2 (HER2) expression by the Immunohistochemical (IHC) method in pathological samples collected from participants with breast cancer.

DETAILED DESCRIPTION:
For accurate selection of participants who will be treated with anti-HER2, primary crucial thing to do is the right identification of HER2 in breast tumor cells. The advantages and disadvantages of IHC and In-Situ Hybridization (ISH) for the detection of HER2 status is still disputable. It is generally agreed on that HER2 study should be applied on all invasive breast cancer participants. It can be used together with IHC which measures HER2 protein expression or ISH which assesses HER2 gene amplification. With regard to IHC, the inconsistency of sensitivity and specificity of marketed antibodies, differences in interpretation and technical artifacts cause problems in diagnosis on occasion. There is not enough study on reasons which cause the consistence and discrepancies between laboratories in HER2 detection with IHC method.

ELIGIBILITY:
Inclusion Criteria:

Samples that fulfill all of the criteria will be evaluated for the study.

* Samples of women aged greater than or equal to (>/=) 18 and less than (<) 75 years
* Tumor samples already diagnosed based on the IHC score of 0 to +3
* Samples of primary lesions excluding lymph nodes
* 10 percent (%) neutral buffered formalin-fixed and paraffin embedded tissue samples

Exclusion Criteria:

Samples that fulfill any of the criteria below will not be included in the study.

* Non-invasive ductal carcinoma (NOS) samples
* Tru-cut biopsies
* Non-breast cancer pathological samples

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast tissue samples from female participants with a breast cancer diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Turkey (Türkiye) (5):
  - Ankara University Medical Faculty, Ankara
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Ege University Medical Faculty, Izmir
  - Dokuz Eylul University Medical Faculty, Izmir

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 5 trial sites (named as Sites A to E) along with 1 reference site (named as Abroad) participated in this study.
Groups:
- Breast Cancer Pathology Participants: Breast cancer pathology participants were evaluated for a period of 70 days.
Period: Overall Study
Arm/Group | Breast Cancer Pathology Participants
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): All enrolled participants.
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 30
Age, Customized [Number; unit: participants]
  ≥ 18 and < 75 years | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Immunohistochemical (IHC) Evaluation Between Site A and Others (Sites B, C, D and E)
Description: IHC is a staining process performed on fresh/frozen breast cancer tissue. IHC is used to show whether or not the cancer cells have Human Epidermal Growth Receptor (HER2) and/or hormone receptors on their surface. The IHC test gives a score of 0 to 3+ that measures the amount of HER2 receptor protein on the surface of cells in a breast cancer tissue sample. Score 0: cells free from immune staining, score 1 (+): is concluded in the case of stains not completely membranous and which do not surround the membranes regardless of quantity in the cells, or weak stains surrounding the entire membrane in less than 10% of the cells. Score 2 (++): is concluded in the presence of a moderate staining surrounding the cytoplasmic membrane in at least 10%, or strong membranous staining in less than 30% of the invasive carcinoma cells. Score 3 (+++): is concluded where IHC yields strong staining surrounding the entire cytoplasmic membrane in at least 30% of the invasive carcinoma cells.
Time Frame: Up to 70 days
Population: FAS population. Here "number of participants analyzed" included evaluable for the outcome measure and "n" included the number of participants evaluable for the specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 24
percentage of participants
  Site A (0): Site B (0) (n=9) | 16.7
  Site A (0): Site B (1+) (n=9) | 12.5
  Site A (0): Site B (2+) (n=9) | 0.0
  Site A (0): Site B (3+) (n=9) | 8.3
  Site A (1+): Site B (0) (n=6) | 4.2
  Site A (1+): Site B (1+) (n=6) | 12.5
  Site A (1+): Site B (2+) (n=6) | 4.2
  Site A (1+): Site B (3+) (n=6) | 4.2
  Site A (2+): Site B (0) (n=5) | 0.0
  Site A (2+): Site B (1+) (n=5) | 4.2
  Site A (2+): Site B (2+) (n=5) | 8.3
  Site A (2+): Site B (3+) (n=5) | 8.3
  Site A (3+): Site B (0) (n=4) | 0.0
  Site A (3+): Site B (1+) (n=4) | 0.0
  Site A (3+): Site B (2+) (n=4) | 16.7
  Site A (3+): Site B (3+) (n=4) | 0.0
  Site A (0): Site C (0) (n=9) | 20.8

2. Primary Outcome: Kappa Coefficient (K) as a Measure of Agreement Between Site A and Others (Sites B, C, D and E) Concerning the IHC Test of Breast Tissue Samples
Description: Inter-laboratory variation between the sites was assessed using Kappa test, K values were interpreted as follows: a) less than (<) 0: less than chance agreement, b) 0.01-0.20: slight agreement, c) 0.21-0.40: fair agreement, d) 0.41-0.60: moderate agreement, e) 0.61-0.80: substantial agreement, and f) 0.81-0.99: almost perfect agreement.
Time Frame: Up to 70 days
Population: FAS population. Here "number of participants analyzed" included evaluable for the outcome measure.
Measure: Number; unit: kappa coefficient
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 24
kappa coefficient
  Site A: Site B | 0.171
  Site A: Site C | 0.090
  Site A: Site D | -0.148
  Site A: Site E | -0.124
Statistical Analysis 1: Comparison: Breast Cancer Pathology Participants; Site A: Site B variability assessment; Test type: Superiority or Other; p = 0.137, Chi-squared
Statistical Analysis 2: Comparison: Breast Cancer Pathology Participants; Site A: Site C variability assessment; Test type: Superiority or Other; p = 0.454, Chi-squared
Statistical Analysis 3: Comparison: Breast Cancer Pathology Participants; Site A: Site D variability assessment; Test type: Superiority or Other; p = 0.211, Chi-squared
Statistical Analysis 4: Comparison: Breast Cancer Pathology Participants; Site A: Site E variability assessment; Test type: Superiority or Other; p = 0.294, Chi-squared

3. Primary Outcome: Percentage of Participants With IHC Evaluation Between Sites B and Others (Sites C, D and E)
Description: IHC is a staining process performed on fresh/frozen breast cancer tissue. IHC is used to show whether or not the cancer cells have HER2 and/or hormone receptors on their surface. The IHC test gives a score of 0 to 3+ that measures the amount of HER2 receptor protein on the surface of cells in a breast cancer tissue sample. Score 0: cells free from immune staining, score 1 (+): is concluded in the case of stains not completely membranous and which do not surround the membranes regardless of quantity in the cells, or weak stains surrounding the entire membrane in less than 10% of the cells. Score 2 (++): is concluded in the presence of a moderate staining surrounding the cytoplasmic membrane in at least 10%, or strong membranous staining in less than 30% of the invasive carcinoma cells. Score 3 (+++): is concluded where IHC yields strong staining surrounding the entire cytoplasmic membrane in at least 30% of the invasive carcinoma cells.
Time Frame: Up to 70 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 24
percentage of participants
  Site B (0): Site C (0) (n=5) | 12.5
  Site B (0): Site C (1+) (n=5) | 4.2
  Site B (0): Site C (2+) (n=5) | 0.0
  Site B (0): Site C (3+) (n=5) | 4.2
  Site B (1+): Site C (0) (n=7) | 4.2
  Site B (1+): Site C (1+) (n=7) | 12.5
  Site B (1+): Site C (2+) (n=7) | 0.0
  Site B (1+): Site C (3+) (n=7) | 12.5
  Site B (2+): Site C (0) (n=6) | 4.2
  Site B (2+): Site C (1+) (n=6) | 4.2
  Site B (2+): Site C (2+) (n=6) | 16.7
  Site B (2+): Site C (3+) (n=6) | 0.0
  Site B (3+): Site C (0) (n=6) | 8.3
  Site B (3+): Site C (1+) (n=6) | 4.2
  Site B (3+): Site C (2+) (n=6) | 12.5
  Site B (3+): Site C (3+) (n=6) | 0.0
  Site B (0): Site D (0) (n=5) | 4.2
  Site B (0): Site D (1+) (n=5) | 0.0
  Site B (0): Site D (+2) (n=5) | 0.0
  Site B (0): Site D (3+) (n=5) | 16.7
  Site B (1+): Site D (0) (n=7) | 12.5
  Site B (1+): Site D (1+) (n=7) | 8.3
  Site B (1+): Site D (2+) (n=7) | 8.3
  Site B (1+): Site D (3+) (n=7) | 0.0
  Site B (2+): Site D (0) (n=6) | 8.3
  Site B (2+): Site D (1+) (n=6) | 16.7
  Site B (2+): Site D (2+) (n=6) | 0.0
  Site B (2+): Site D (3+) (n=6) | 0.0
  Site B (3+): Site D (0) (n=6) | 4.2
  Site B (3+): Site D (1+) (n=6) | 4.2
  Site B (3+): Site D (2+) (n=6) | 4.2
  Site B (3+): Site D (3+) (n=6) | 12.5
  Site B (0): Site E (0) (n=5) | 12.5
  Site B (0): Site E (1+) (n=5) | 4.2
  Site B (0): Site E (2+) (n=5) | 4.2
  Site B (0): Site E (3+) (n=5) | 0.0
  Site B (1+): Site E (0) (n=7) | 0.0
  Site B (1+): Site E (1+) (n=7) | 0.0
  Site B (1+): Site E (2+) (n=7) | 8.3
  Site B (1+): Site E (3+) (n=7) | 20.8
  Site B (2+): Site E (0) (n=6) | 8.3
  Site B (2+): Site E (1+) (n=6) | 4.2
  Site B (2+): Site E (2+) (n=6) | 12.5
  Site B (2+): Site E (3+) (n=6) | 0.0
  Site B (3+): Site E (0) (n=6) | 8.3
  Site B (3+): Site E (1+) (n=6) | 12.5
  Site B (3+): Site E (2+) (n=6) | 4.2
  Site B (3+): Site E (3+) (n=6) | 0.0

4. Primary Outcome: Kappa Coefficient as a Measure of Agreement Between Site B and Others (Sites C, D and E) Concerning the IHC Test of Breast Tissue Samples
Description: Inter-laboratory variation between the sites was assessed using Kappa test, K values to be interpreted as follows: a) <0: less than chance agreement, b) 0.01-0.20: slight agreement, c) 0.21-0.40: fair agreement, d) 0.41-0.60: moderate agreement, e) 0.61-0.80: substantial agreement, and f) 0.81-0.99: almost perfect agreement.
Time Frame: Up to 70 days
Population: FAS population. Here "number of participants analyzed" included evaluable for the outcome measure.
Measure: Number; unit: kappa coefficient
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 24
kappa coefficient
  Site B: Site C | 0.224
  Site B: Site D | 0.000
  Site B: Site E | 0.05
Statistical Analysis 1: Comparison: Breast Cancer Pathology Participants; Site B: Site C variability assessment; Test type: Superiority or Other; p = 0.054, Chi-squared
Statistical Analysis 2: Comparison: Breast Cancer Pathology Participants; Site B: Site D variability assessment; Test type: Superiority or Other; p = 1.000, Chi-squared
Statistical Analysis 3: Comparison: Breast Cancer Pathology Participants; Site B: Site E variability assessment; Test type: Superiority or Other; p = 0.968, Chi-squared

5. Secondary Outcome: Percentage of Participants With Diagnosis of Primary Tumor
Description: Primary tumor diagnosis was classified into invasive ductal carcinoma, invasive ductal carcinoma + integrin linked kinase (ILK) antibody and mixed (invasive ductal + lobular) and reported.
Time Frame: Up to 70 days
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 30
percentage of participants
  Invasive ductal carcinoma | 93.3
  Invasive ductal carcinoma + ILK | 3.3
  Mixed (Invasive Ductal+Lobular) | 3.3

6. Secondary Outcome: Percentage of Participants With Initial Tumor Node Metastasis (TNM) Stage According to Council Decision
Description: TNM system is based on size of primary tumor (T), amount of spread to lymph nodes (N) and presence of metastasis (M). T1: tumor ≤20 millimeters (mm), T2: tumor >20 mm to ≤50 mm, T3: >50 mm and TX: tumor cannot be assessed. N0: no lymph node metastasis, N1: metastasis to ipsilateral level I, II axillary lymph nodes, N2: N1 metastasis that is clinically fixed/matted or in clinically detected ipsilateral internal mammary nodes, N3: metastases in ipsilateral infraclavicular lymph nodes, with/without level I, II axillary node involvement, or in clinically detected ipsilateral internal mammary lymph nodes and clinically evident level I, II axillary lymph node metastasis; or metastasis in ipsilateral supraclavicular lymph nodes, NX: Regional lymph nodes cannot be assessed. M0: no clinical/radiographic evidence of distant metastasis, M1: distant detectable metastases as determined by clinical and radiographic means and/or histologically proven >0.2 mm, and MX: metastases cannot be assessed.
Time Frame: Up to 70 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 24
percentage of participants
  T1 (n=24) | 33.3
  T2 (n=24) | 54.2
  T3 (n=24) | 8.3
  TX (n=24) | 4.2
  N0 (n=24) | 50.0
  N1 (n=24) | 16.7
  N2 (n=24) | 20.8
  N3 (n=24) | 8.3
  NX (n=24) | 4.2
  M0 (n=18) | 50.0
  M1 (n=18) | 11.1
  MX (n=18) | 38.9

7. Secondary Outcome: Percentage of Participants With Pathological Score
Description: Modified Bloom-Richardson Grade scoring system was used which considers the amount of glandular/tubular differentiation, nuclear features and the mitotic activity of tumor cells. Tubular score (TS) 1: >75 percent (%) of tumor area forming tubular structures, TS 2: 10% to 75% of tumor area forming tubular structures, TS 3: <10% of tumor area forming tubular structures. Nuclear score (NS) 1: nuclei small with little increase in size in comparison with normal breast epithelial cells, regular outlines, uniform nuclear chromatin, little variation in size, NS 2: cells larger than normal with open vesicular nuclei, visible nucleoli, and moderate variability in both size and shape, NS 3: Vesicular nuclei, often with prominent nucleoli, exhibiting marked variation in size and shape, occasionally with very large and bizarre forms. Mitosis score (MS) 1: ≤7 mitoses per 10 high power fields, MS 2: 8-14 mitoses per 10 high power fields and MS 3: ≥15 mitoses per 10 high power fields.
Time Frame: Up to 70 days
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 30
percentage of participants
  TS 1 | 0.0
  TS 2 | 43.3
  TS 3 | 56.7
  NS 1 | 0.0
  NS 2 | 33.3
  NS 3 | 66.7
  MS 1 | 20.0
  MS 2 | 63.3
  MS 3 | 16.7

8. Secondary Outcome: Percentage of Participants With Pathological Grade
Description: Modified Bloom-Richardson Grade scoring system was used which considers the amount of glandular/tubular differentiation, nuclear features and the mitotic activity of tumor cells. Tubular, Nuclear and Mitosis scoring pattern was discussed in outcome 11, each score was added to give a final total score ranging from 3-9. Tumors with 3, 4 or 5 points are classified as being of low malignancy or Grade I, those with 6 or 7 points of intermediate malignancy or Grade II, and those with 8 or 9 points of high malignancy or Grade III.
Time Frame: Up to 70 days
Population: FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 30
percentage of participants
  Grade I Tumor | 0.0
  Grade II Tumor | 56.7
  Grade III Tumor | 43.3

9. Secondary Outcome: Percentage of Participants With Different Hormone Receptors
Description: Presence of hormone receptors was examined by the amount of uptake of estrogen and progesterone hormones when analyzed using IHC staining procedure.
Time Frame: Up to 70 days
Population: FAS population. Here "number of participants analyzed" included evaluable for the outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 27
percentage of participants
  Estrogen receptors | 71.3
  Progesterone receptors | 42.69

10. Secondary Outcome: Percentage of Participants With Specified Density of Hormone Receptors
Description: The specific density of hormone receptors was examined by the amount of uptake of estrogen and progesterone hormones when analyzed using IHC staining procedure. Score 0: cells free from immune staining, score 1 (+): is concluded in the case of stains not completely membranous and which do not surround the membranes regardless of quantity in the cells, or weak stains surrounding the entire membrane in less than 10% of the cells. Score 2 (++): is concluded in the presence of a moderate staining surrounding the cytoplasmic membrane in at least 10%, or strong membranous staining in less than 30% of the invasive carcinoma cells. Score 3 (+++): is concluded where IHC yields strong staining surrounding the entire cytoplasmic membrane in at least 30% of the invasive carcinoma cells.
Time Frame: Up to 70 days
Population: FAS population. Here "number of participants analyzed" included evaluable for the outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 25
percentage of participants
  Estrogen receptor density unknown | 4.0
  Estrogen receptor density + | 8.0
  Estrogen receptor density ++ | 16.0
  Estrogen receptor density +++ | 72.0
  Progesterone receptor density 0 | 12.0
  Progesterone receptor density ++ | 28.0
  Progesterone receptor density +++ | 60.0

11. Secondary Outcome: Percentage of Participants With HER2 Test Form Based on Country
Description: Reference site was considered as Abroad and the tests were performed in a laboratory in Amsterdam, Netherlands. A total of 150 data registration forms (120 forms from trial sites [24 from each site] and 30 from the reference site) were collected.
Time Frame: Up to 70 days
Population: FAS population.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Data registration forms
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 30
Number analyzed (Data registration forms) | 150
percentage of participants
  Turkey | 80.0
  Abroad | 20.0

12. Secondary Outcome: Percentage of Participants With HER2 Test Form Based on Different Automated Slide Stainers
Description: Different slide stainers like Ventana, Ventana Benchmark 4XT, Ventana Benchmark Ultra and Ventana Benchmark XT were used to report HER2 test results on data registration forms (120 forms from trial sites [24 from each site] and 30 from the reference site).
Time Frame: Up to 70 days
Population: FAS population.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Data registration forms
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 30
Number analyzed (Data registration forms) | 150
percentage of participants
  Ventana | 20.0
  Ventana Benchmark 4XT | 16.0
  Ventana Benchmark Ultra | 16.0
  Ventana Benchmark XT | 48.0

13. Secondary Outcome: Percentage of Participants With HER2 Test Form Based on Antigen Retrieval
Description: Fixation of tissue samples cross-link proteins and masks antigenic sites; antigen retrieval process was performed before IHC staining in order to reverse the masking of antigenic sites. Antigen retrieval process was performed in this study using the following solutions: 1 hour Cell Conditioning 1 (CC1), 30 minutes (min) CC1 mild, 64 min CC1, CC1 Ethylenediaminetetraacetic acid (EDTA) standard, and Cell Conditioning 2 (CC2) 30 min.
Time Frame: Up to 70 days
Population: FAS population.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Data registration forms
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 30
Number analyzed (Data registration forms) | 150
percentage of participants
  1 hour CC1 | 16.0
  30 min CC1 mild | 32.0
  64 min CC1 | 16.0
  CC1 EDTA standard | 16.0
  CC2 30 min | 20.0

14. Secondary Outcome: Percentage of Participants With HER2 Test Form Based on Primary Antibody
Description: The primary antibodies included; Biocabe EP 10454, Cerb B2 (SP3 clone), Her2 Neu (SP3) Cell marque, Neomarkers (thermo) cerb B2-Ab-17 and Thermo SP3.
Time Frame: Up to 70 days
Population: FAS population.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Data registration forms
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 30
Number analyzed (Data registration forms) | 150
percentage of participants
  Biocabe EP 10454 | 16.0
  Cerb B2 (SP3 clone) | 16.0
  Her2 Neu (SP3) Cell marque | 16.0
  Neomarkers (thermo) cerb B2-Ab-17 | 16.0
  Thermo SP3 | 36.0

15. Secondary Outcome: Percentage of Participants With Different IHC Results
Description: The IHC test gives a score of 0 to 3+ that measures the amount of HER2 receptor protein on the surface of cells in a breast cancer tissue sample. If the score is 0 to 1+, it's called "HER2 negative." If the score is 2+, it's called "borderline." A score of 3+ is called "HER2 positive." Score 0: cells free from immune staining, score 1 (+): is concluded in the case of stains not completely membranous and which do not surround the membranes regardless of quantity in the cells, or weak stains surrounding the entire membrane in less than 10% of the cells. Score 2 (++): is concluded in the presence of a moderate staining surrounding the cytoplasmic membrane in at least 10%, or strong membranous staining in less than 30% of the invasive carcinoma cells. Score 3 (+++): is concluded where IHC yields strong staining surrounding the entire cytoplasmic membrane in at least 30% of the invasive carcinoma cells.
Time Frame: Up to 70 days
Population: FAS population.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Data registration forms
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 30
Number analyzed (Data registration forms) | 150
percentage of participants
  IHC 0 | 36.7
  IHC 1+ | 20.7
  IHC 2+ | 20.7
  IHC 3+ | 22.0

16. Primary Outcome: Percentage of Participants With IHC Evaluation Between Site C and Others (Sites D and E)
Description: as for outcome 3
Time Frame: Up to 70 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 24
percentage of participants
  Site C (0): Site D (0) (n=9) | 8.3
  Site C (0): Site D (1+) (n=9) | 4.2
  Site C (0): Site D (2+) (n=9) | 8.3
  Site C (0): Site D (3+) (n=9) | 16.7
  Site C (1+): Site D (0) (n=5) | 4.2
  Site C (1+): Site D (1+) (n=5) | 4.2
  Site C (1+): Site D (2+) (n=5) | 4.2
  Site C (1+): Site D (3+) (n=5) | 12.5
  Site C (2+): Site D (0) (n=6) | 8.3
  Site C (2+): Site D (1+) (n=6) | 12.5
  Site C (2+): Site D (2+) (n=6) | 4.2
  Site C (2+): Site D (3+) (n=6) | 0.0
  Site C (3+): Site D (0) (n=4) | 16.7
  Site C (3+): Site D (1+) (n=4) | 0.0
  Site C (3+): Site D (2+) (n=4) | 0.0
  Site C (3+): Site D (3+) (n=4) | 0.0
  Site C (0): Site E (0) (n=9) | 25.0
  Site C (0): Site E (1+) (n=9) | 4.2
  Site C (0): Site E (2+) (n=9) | 0.0
  Site C (0): Site E (3+) (n=9) | 8.3
  Site C (1+): Site E (0) (n=5) | 4.2
  Site C (1+): Site E (1+) (n=5) | 8.3
  Site C (1+): Site E (2+) (n=5) | 0.0
  Site C (1+): Site E (3+) (n=5) | 8.3
  Site C (2+): Site E (0) (n=6) | 4.2
  Site C (2+): Site E (1+) (n=6) | 8.3
  Site C (2+): Site E (2+) (n=6) | 12.5
  Site C (2+): Site E (3+) (n=6) | 0.0
  Site C (3+): Site E (0) (n=4) | 0.0
  Site C (3+): Site E (1+) (n=4) | 0.0
  Site C (3+): Site E (2+) (n=4) | 16.7
  Site C (3+): Site E (3+) (n=4) | 0.0
  Site D (0): Site E (0) (n=10) | 4.2
  Site D (0): Site E (1+) (n=10) | 12.5
  Site D (0): Site E (2+) (n=10) | 16.7
  Site D (0): Site E (3+) (n=10) | 8.3
  Site D (1+): Site E (0) (n=5) | 8.3
  Site D (1+): Site E (1+) (n=5) | 0.0
  Site D (1+): Site E (2+) (n=5) | 4.2
  Site D (1+): Site E (3+) (n=5) | 8.3
  Site D (2+): Site E (0) (n=2) | 4.2
  Site D (2+): Site E (1+) (n=2) | 0.0
  Site D (2+): Site E (2+) (n=2) | 0.0
  Site D (2+): Site E (3+) (n=2) | 4.2
  Site D (3+): Site E (0) (n=7) | 20.8
  Site D (3+): Site E (1+) (n=7) | 4.2
  Site D (3+): Site E (2+) (n=7) | 4.2
  Site D (3+): Site E (3+) (n=7) | 0.0

17. Primary Outcome: Kappa Coefficient as a Measure of Agreement Between Sites C, D and E Concerning the IHC Test of Breast Tissue Samples
Description: as for outcome 4
Time Frame: Up to 70 days
Population: FAS population. Here "number of participants analyzed" included evaluable for the outcome measure.
Measure: Number; unit: kappa coefficient
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 24
kappa coefficient
  Site C: Site D | -0.137
  Site C: Site E | 0.259
  Site D: Site E | -0.317
Statistical Analysis 1: Comparison: Breast Cancer Pathology Participants; Site C: Site D variability assessment; Test type: Superiority or Other; p = 0.246, Chi-squared
Statistical Analysis 2: Comparison: Breast Cancer Pathology Participants; Site C: Site E variability assessment; Test type: Superiority or Other; p = 0.032, Chi-squared
Statistical Analysis 3: Comparison: Breast Cancer Pathology Participants; Site D: Site E variability assessment; Test type: Superiority or Other; p = 0.007, Chi-squared

18. Primary Outcome: Percentage of Participants With IHC Evaluation Between Abroad and Trial Sites (A, B, C, D and E)
Description: as for outcome 3
Time Frame: Up to 70 days
Population: FAS population. "n" included the number of participants evaluable for the specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 30
percentage of participants
  Abroad (0): Site A (0) (n=13) | 16.7
  Abroad (0): Site A (1+) (n=13) | 13.3
  Abroad (0): Site A (2+) (n=13) | 10.0
  Abroad (0): Site A (3+) (n=13) | 3.3
  Abroad (1+): Site A (0) (n=4) | 6.7
  Abroad (1+): Site A (1+) (n=4) | 3.3
  Abroad (1+): Site A (2+) (n=4) | 3.3
  Abroad (1+): Site A (3+) (n=4) | 0.0
  Abroad (2+): Site A (0) (n=6) | 0.0
  Abroad (2+): Site A (1+) (n=6) | 6.7
  Abroad (2+): Site A (2+) (n=6) | 3.3
  Abroad (2+): Site A (3+) (n=6) | 10.0
  Abroad (3+): Site A (0) (n=7) | 10.0
  Abroad (3+): Site A (1+) (n=7) | 3.3
  Abroad (3+): Site A (2+) (n=7) | 6.7
  Abroad (3+): Site A (3+) (n=7) | 3.3
  Abroad (0): Site B (0) (n=13) | 13.3
  Abroad (0): Site B (1+) (n=13) | 13.3
  Abroad (0): Site B (2+) (n=13) | 6.7
  Abroad (0): Site B (3+) (n=13) | 10.0
  Abroad (1+): Site B (0) (n=4) | 3.3
  Abroad (1+): Site B (1+) (n=4) | 6.7
  Abroad (1+): Site B (2+) (n=4) | 3.3
  Abroad (1+): Site B (3+) (n=4) | 0.0
  Abroad (2+): Site B (0) (n=6) | 0.0
  Abroad (2+): Site B (1+) (n=6) | 3.3
  Abroad (2+): Site B (2+) (n=6) | 13.3
  Abroad (2+): Site B (3+) (n=6) | 3.3
  Abroad (3+): Site B (0) (n=7) | 3.3
  Abroad (3+): Site B (1+) (n=7) | 6.7
  Abroad (3+): Site B (2+) (n=7) | 3.3
  Abroad (3+): Site B (3+) (n=7) | 10.0
  Abroad (0): Site C (0) (n=13) | 20.0
  Abroad (0): Site C (1+) (n=13) | 10.0
  Abroad (0): Site C (2+) (n=13) | 6.7
  Abroad (0): Site C (3+) (n=13) | 6.7
  Abroad (1+): Site C (0) (n=4) | 3.3
  Abroad (1+): Site C (1+) (n=4) | 6.7
  Abroad (1+): Site C (2+) (n=4) | 0.0
  Abroad (1+): Site C (3+) (n=4) | 3.3
  Abroad (2+): Site C (0) (n=6) | 0.0
  Abroad (2+: Site C (1+) (n=6) | 3.3
  Abroad (2+): Site C (2+) (n=6) | 13.3
  Abroad (2+): Site C (3+) (n=6) | 3.3
  Abroad (3+): Site C (0) (n=7) | 10.0
  Abroad (3+): Site C (1+) (n=7) | 3.3
  Abroad (3+): Site C (2+) (n=7) | 6.7
  Abroad (3+): Site C (3+) (n=7) | 3.3
  Abroad (0): Site D (0) (n=13) | 10.0
  Abroad (0): Site D (1+) (n=13) | 13.3
  Abroad (0): Site D (2+) (n=13) | 3.3
  Abroad (0): Site D (3+) (n=13) | 16.7
  Abroad (1+): Site D (0) (n=4) | 6.7
  Abroad (1+): Site D (1+) (n=4) | 3.3
  Abroad (1+): Site D (2+) (n=4) | 3.3
  Abroad (1+): Site D (3+) (n=4) | 0.0
  Abroad (2+): Site D (0) (n=6) | 16.7
  Abroad (2+): Site D (1+) (n=6) | 3.3
  Abroad (2+): Site D (2+) (n=6) | 0.0
  Abroad (2+): Site D (3+) (n=6) | 0.0
  Abroad (3+): Site D (0) (n=7) | 3.3
  Abroad (3+): Site D (1+) (n=7) | 3.3
  Abroad (3+): Site D (2+) (n=7) | 6.6
  Abroad (3+): Site D (3+) (n=7) | 9.9
  Abroad (0): Site E (0) (n=13) | 16.7
  Abroad (0): Site E (1+) (n=13) | 6.7
  Abroad (0): Site E (2+) (n=13) | 13.3
  Abroad (0): Site E (3+) (n=13) | 6.7
  Abroad (1+): Site E (0) (n=4) | 3.3
  Abroad (1+): Site E (1+) (n=4) | 0.0
  Abroad (1+): Site E (2+) (n=4) | 3.3
  Abroad (1+): Site E (3+) (n=4) | 6.7
  Abroad (2+): Site E (0) (n=6) | 6.7
  Abroad (2+): Site E (1+) (n=6) | 6.7
  Abroad (2+): Site E (2+) (n=6) | 6.7
  Abroad (2+): Site E (3+) (n=6) | 0.0
  Abroad (3+): Site E (0) (n=7) | 6.7
  Abroad (3+): Site E (1+) (n=7) | 6.7
  Abroad (3+): Site E (2+) (n=7) | 3.3
  Abroad (3+): Site E (3+) (n=7) | 6.7

19. Primary Outcome: Kappa Coefficient as a Measure of Agreement Between Abroad and Trial Sites (A, B, C, D and E) Concerning the IHC Test of Breast Tissue Samples
Description: as for outcome 4
Time Frame: Up to 70 days
Population: FAS population.
Measure: Number; unit: kappa coefficient
Arm/Group | Breast Cancer Pathology Participants
Number analyzed (Participants) | 30
kappa coefficient
  Abroad: Site A | 0.002
  Abroad: Site B | 0.260
  Abroad: Site C | 0.226
  Abroad: Site D | -0.063
  Abroad: Site E | 0.04
Statistical Analysis 1: Comparison: Breast Cancer Pathology Participants; Abroad: Site A variability assessment; Test type: Superiority or Other; p = 0.988, Chi-squared
Statistical Analysis 2: Comparison: Breast Cancer Pathology Participants; Abroad: Site B variability assessment; Test type: Superiority or Other; p = 0.008, Chi-squared
Statistical Analysis 3: Comparison: Breast Cancer Pathology Participants; Abroad: Site C variability assessment; Test type: Superiority or Other; p = 0.031, Chi-squared
Statistical Analysis 4: Comparison: Breast Cancer Pathology Participants; Abroad: Site D variability assessment; Test type: Superiority or Other; p = 0.554, Chi-squared
Statistical Analysis 5: Comparison: Breast Cancer Pathology Participants; Abroad: Site E variability assessment; Test type: Superiority or Other; p = 0.709, Chi-squared

ADVERSE EVENTS:
Description: As the present study was non-interventional and performed on biology samples obtained from participants, it was not planned to collect adverse events data.
Arm/Group | Breast Cancer Pathology Participants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.